CLINICAL TRIAL: NCT02692352
Title: Cognitive Rehabilitation of Executive Dysfunction - Goal Management Training in Patients With Acquired Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: University of Oslo (Other); University of Glasgow (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Sveinung Tornaas, Principal investigator, Sunnaas Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011/2/0204
Record Dates: First submitted 2016-02-23; First posted 2016-02-26 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): 8 sessions of Goal Management Training
  Interventions: Other: Goal Management Training
- Active control group (Active Comparator): 8 sessions of Brain Health Workshop
  Interventions: Other: Brain Health Workshop

INTERVENTIONS:
Other: Goal Management Training — Goal Management training, 8 sessions of 2 hours
  Arms: Experimental
Other: Brain Health Workshop — Brain Health Workshop training, 8 sessions of 2 hours
  Arms: Active control group

SUMMARY:
The main objective of this study is to examine the effect of Goal Management Training for patients with executive difficulties after acquired brain injury in a randomized controlled trial. The effect on cognitive functioning will be examined, as will the relationship between treatment effects and lesion location and size. The effect of Goal Management training on regulating emotions, quality of life and coping will be examined. The generalizability of treatment effects across etiologies will be explored by comparing effects in three patient groups; traumatic brain injury, cerebrovascular accidents and resected brain tumors. Structural Magnetic Resonance Imaging (MRI) scans and measures of white matter connectivity will be used to establish detailed lesion descriptions. Functional MRI data will provide information on the neural underpinnings of treatment related change. A secondary objective is to expand the Goal Management Training protocol with increased focus on emotional regulation and adherence to homework assignment.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic Brain Injury, stroke and resected brain tumor patients with no concomitant diseases
* Minimum 6 months post-injury/surgery
* Reporting executive problems by structured interview or baseline assessment (cognitive performance measures)

Exclusion Criteria:

* Major psychiatric disorder or reported ongoing alcohol or substance abuse
* Premorbid neurological disease or insult and/or comorbid neurological disease
* Aphasia or other specified language problems causing potential communication problems
* Impaired basic cognitive, linguistic, mnemonic, motor, or perceptual function that can interfere with the ability to engage with the training

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Executive functioning in daily life measured by self report questionnaire | one year
  Behavior Rating Inventory Executive Functions Adult version
Executive functioning measured by neuropsychological assessment | one year
  Conners Continous Performance Test

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olsen A, Dennis EL, Stubberud J, Hovenden ES, Solbakk AK, Endestad T, Kristian Hol P, Schanke AK, Lovstad M, Tornas S. Regional brain volume prior to treatment is linked to outcome after cognitive rehabilitation in traumatic brain injury. Neuroimage Clin. 2022;35:103126. doi: 10.1016/j.nicl.2022.103126. Epub 2022 Jul 28. PMID 36002956
- [Derived] Tornas S, Lovstad M, Solbakk AK, Schanke AK, Stubberud J. Goal Management Training Combined With External Cuing as a Means to Improve Emotional Regulation, Psychological Functioning, and Quality of Life in Patients With Acquired Brain Injury: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2016 Nov;97(11):1841-1852.e3. doi: 10.1016/j.apmr.2016.06.014. Epub 2016 Jul 15. PMID 27424292